CLINICAL TRIAL: NCT01376713
Title: CD20-Immunotargeting in Metastatic Melanoma Patients- A Prospective, Open Label, Sequential Pilot Study
Brief Title: Anti-CD20 (Cluster of Differentiation Antigen 20) Therapy to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephan N. Wagner, MD, MD, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2010-023277-19
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Stage III Melanoma; Stage IV Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — ofatumumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ofatumumab alone (Experimental): Patients with melanoma unresectable stage III B (T1- 4a, N2b-c), stage III C or stage IV (AJCC 2009) will be included in this study. Ofatumumab will be administered at a dose of 1000mg iv weekly for 8 weeks and q4w for another 16 weeks. Tumor imaging is performed at wk 4 (screening for rapid disease progression), 8, 16 and 24. In case of PD, patients will have the opportunity to receive at least 3 cycles of ofatumumab q4w in combination with DTIC (1000 mg/m2) q4w (see Arm2).
  Interventions: Biological: Ofatumumab
- Ofatumumab plus Dacarbazine (Experimental): Patients will be treated with a combination of DTIC (1000 mg/m2) q4w plus ofatumumab (1000mg) qw for 8 wks, and thereafter q4w.Tumor imaging is performed at wk 8, 16 and 24.
  Interventions: Biological: Ofatumumab plus Dacarbazine

INTERVENTIONS:
Biological: Ofatumumab — Ofatumumab will be administered at a dose of 1000mg iv weekly for 8 weeks and q4w for another 16 weeks
  Other Names: Arzerra
  Arms: Ofatumumab alone
Biological: Ofatumumab plus Dacarbazine — Ofatumumab will be administered at a dose of 1000mg iv weekly for 8 weeks and q4w for another 16 weeks.
  Dacarbazine administered q4w at a dose of 1000mg/m2, 4 days before next administration of Ofatumumab for 24 weeks.
  Other Names: Arzerra; DTIC
  Arms: Ofatumumab plus Dacarbazine

SUMMARY:
The purpose of this study is to assess the overall disease control rate of Ofatumumab wo/w Dacarbazine in subjects with American Joint Committee on Cancer (AJCC 2009) unresectable stage III or stage IV melanoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, sequential, 2-cohort, phase 2 study to assess the overall disease control rate of Ofatumumab according to criteria of RECIST (Response Evaluation Criteria in Solid Tumors) v. 1.1. in subjects with unresectable stage III B (T1- 4a, N2b-c), stage III C or stage IV (American Joint Committee on Cancer 2009) disease.

Cohort 1: 10 eligible patients will be treated with ofatumumab alone. If interim analysis shows that at least 1 confirmed overall response occurs, an additional 19 eligible patients will be treated, for a total of 29 patients.

Cohort 2: If no confirmed overall response by ofatumumab alone-therapy is seen in the first 10 patients, cohort 2 will be opened. Initially, 13 eligible patients will be treated with a combination of Dacarbazine plus ofatumumab. If interim analysis gives at least 2 confirmed overall responses, additional 26 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Signed informed consent
* Metastatic non-ocular melanoma - unresectable stage III B (T1- 4a, N2b-c), stage III C (AJCC 2009) or stage IV (AJCC 2009).
* measurable disease with more than one metastatic lesion, according to RECIST v. 1.1 criteria,
* One of these metastases must be resectable prior to anti-CD20 therapy.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
* As soon as BRAF or other kinase inhibitors are standard of care, we will include only patients who cannot be considered for those therapies. E.g. patients with tumors not carrying the respective mutational profile, patients refusing this kind of therapy for any reason, patients being not eligible to those therapies due to contraindications or disease progression under such kind of therapy.
* Life expectancy of 3 month or longer
* Negative pregnancy test in female patients of childbearing potential and adequate contraception in female patients of childbearing age.

Exclusion Criteria:

* Patients with active brain metastasis (exception: brain metastases being stable with and without corticosteroids for 2 months after treatment by surgery or radiation therapy) and immunoglobulin-deficiency will be excluded.

Subjects meeting any of the following criteria must not be enrolled in an ofatumumab study:

* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* HIV positive
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to enrollment, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb (HC antibodies), in which case reflexively perform a HC RIBA (recombinant immunoblot assay) on the same sample to confirm the result
* Screening laboratory values:

hemoglobin < 8g/dL platelets <70 x 109/L leukocytes <1.5 x 109/L creatinine >2.0 times ULN (upper limit of normal) total bilirubin >1.5 times ULN liver transaminase ALT >2.5 times ULN alkaline phosphatase >2.5 times ULN

* Pregnant or lactating women
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Disease control according to RECIST v. 1.1 criteria | 24 weeks
  Disease control according to RECIST v. 1.1 criteria until week 24

SECONDARY OUTCOMES:
Assessment of progression-free survival (PFS) | approximately 2 years
  Assessment of progression-free survival (PFS) defined as the time from first day of treatment to the first documentation of disease progression or death, whichever occurs first.
Evaluation of cell biological responses | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
  in patients' blood and tumor samples
Duration of disease control | approximately 2 years
Overall survival | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephan N Wagner, MD, Principal Investigator — Medical University of Vienna; Klemens Rappersberger, Prof. Dr., Principal Investigator — Hospital Rudolfstiftung
Locations (2):
- Austria (2):
  - Rudolfstiftung, Vienna
  - Medical University of Vienna, Vienna

REFERENCES:
- [Background] Balch CM, Gershenwald JE, Soong SJ, Thompson JF, Atkins MB, Byrd DR, Buzaid AC, Cochran AJ, Coit DG, Ding S, Eggermont AM, Flaherty KT, Gimotty PA, Kirkwood JM, McMasters KM, Mihm MC Jr, Morton DL, Ross MI, Sober AJ, Sondak VK. Final version of 2009 AJCC melanoma staging and classification. J Clin Oncol. 2009 Dec 20;27(36):6199-206. doi: 10.1200/JCO.2009.23.4799. Epub 2009 Nov 16. PMID 19917835